CLINICAL TRIAL: NCT01682863
Title: A Multi-centre Randomized Double Blind 52-week Study to Assess the Safety of QVA149 Compared to QAB149 in Patients With COPD Who Have Moderate to Severe Airflow Limitation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149A2340; 2012-001998-93
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, QAB149, QVA149, indacaterol maleate, gylcopyrronium bromide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- QVA149 dose 1 (Experimental): QVA149 27.5/12.5 μg capsules
  Interventions: Drug: QVA149
- QVA149 dose 2 (Experimental): QVA149 27.5/25 μg capsules
  Interventions: Drug: QVA149
- QAB149 (Active Comparator): QAB149 75 μg capsules
  Interventions: Drug: QAB149; Drug: Placebo

INTERVENTIONS:
Drug: QVA149 — QVA149 will be supplied in a capsule form in blister packs for use in the Novartis Concept1 SDDPI
  Arms: QVA149 dose 1
Drug: QVA149 — QVA149 will be supplied in a capsule form in blister packs for use in the Novartis Concept1 SDDPI
  Arms: QVA149 dose 2
Drug: QAB149 — QAB149 and matching placebo will be supplied in capsule form in blister packs for use in the Novartis Concept1 SDDPI
  Arms: QAB149
Drug: Placebo — To mimic QAB149
  Arms: QAB149

SUMMARY:
This study is to assess the safety and tolerability of two different doses of QVA149 and QAB149 in patients with moderate to severe airflow limitation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥40 years
* Patients with stable COPD according to GOLD strategy (GOLD 2011).
* Patients with airflow limitation indicated by a post-bronchodilator FEV1 ≥ 30% and <80% of the predicted normal, and a post-bronchodilator FEV1/FVC < 0.70.
* Current or ex-smokers who have a smoking history of at least 10 pack years.
* Patients with an mMRC ≥ grade 2

Exclusion Criteria:

* History of long QT syndrome or prolonged QTc
* Patients who have had a COPD exacerbation that required treatment with antibiotics and/or systemic corticosteroids and/or hospitalization in the 6 weeks prior to Visit 1.
* Patients with Type I or uncontrolled Type II diabetes
* Patients with a history of asthma or have concomitant pulmonary disease
* Patients with paroxysmal (e.g. intermittent) atrial fibrillation. Only patients with persistent atrial fibrillation and controlled with a rate control strategy for at least six months could be eligible
* Patients who have clinically significant renal, cardiovascular, neurological, endocrine, immunological, psychiatric, gastrointestinal, hepatic, or hematological abnormalities which could interfere with the assessment of safety
* Other protocol defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (80):
- United States (46):
  - Novartis Investigative Site, Vestavia Hills, Alabama
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Lakewood, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Lombard, Illinois
  - Novartis Investigative Site, O'Fallon, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Ames, Iowa
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Waterloo, Iowa
  - Novartis Investigative Site, Bowling Green, Kentucky
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Livonia, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Dublin, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Corsicana, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Lufkin, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, Abingdon, Virginia
  - Novartis Investigative Site, Midlothian, Virginia
  - Novartis Investigative Site, Newport News, Virginia
- Bulgaria (5):
  - Novartis Investigative Site, Rousse, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Varna, Bulgaria
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
- Finland (4):
  - Novartis Investigative Site, Helsinki, Finland
  - Novartis Investigative Site, HUS
  - Novartis Investigative Site, Pori
  - Novartis Investigative Site, Turku
- Hungary (8):
  - Novartis Investigative Site, Nyíregyháza, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Százhalombatta
  - Novartis Investigative Site, Szolnok
  - Novartis Investigative Site, Törökbálint
- Puerto Rico (2):
  - Novartis Investigative Site, Barceloneta
  - Novartis Investigative Site, San Juan
- Romania (7):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Constanța, Jud. Constanta
  - Novartis Investigative Site, Iași, Jud. Iasi
  - Novartis Investigative Site, Brasov, Romania
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Spain (8):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Canet de Mar, Catalonia
  - Novartis Investigative Site, Centelles, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to each treatment arm in 1:1:1 ratio.
Pre-assignment Details: Six hundred fifteen patients were randomized. One patient was randomized but did not receive treatment due to an adverse event. In the safety set, patients were analyzed according to the treatment received. Therefore, protocol enrollment and analysis set was 614 but the participant flow was 615
Period: Overall Study
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od
Started | 204 | 204 | 207
Safety Set | 204 | 204 | 206
Full Analysis Set (FAS) | 204 (included all randomized patients who received at least one dose of study medication) | 204 | 206
Randomized Set | 204 | 204 | 207 (1 randomized patient was not treated; experienced an AE prior to receiving any study drug)
Completed | 177 | 187 | 183
Not Completed | 27 | 17 | 24
Not completed — Subject/guardian decision | 19 | 12 | 10
Not completed — Lost to Follow-up | 5 | 1 | 6
Not completed — Death | 1 | 3 | 4
Not completed — Protocol deviation | 1 | 0 | 1
Not completed — Technical problems | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis set (FAS) included all randomized patients who received at least one dose of study medication. Patients were analyzed according to the treatment they were assigned to at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od | Total
Number analyzed (Participants) | 204 | 204 | 207 | 615
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (7.90) | 63.9 (8.50) | 62.8 (8.52) | 63.6 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 81 | 58 | 212
  Male | 131 | 123 | 149 | 403

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events, Serious Adverse Events, and Death
Description: The overall rate of adverse events reported from initiation through 30 days post last dose.
Time Frame: 56 weeks
Population: The Safety set:all patients that received at least one dose of study medication and had at least one post-baseline safety assessment. Patients were analyzed according to treatment received. The statement that a patient had no AEs also constituted a safety assessment. Only deaths occurring on treatment + 30 days after end of treatment were included.
Measure: Number; unit: Number of Patients
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od
Number analyzed (Participants) | 204 | 204 | 206
Number of Patients
  Patients with at least one SAEs | 26 | 25 | 24
  Patients with at least one AE | 139 | 142 | 139
  Death | 1 | 3 | 5

2. Secondary Outcome: Time to Premature Discontinuation of Treatment
Description: methodTime to premature treatment discontinuation for each treatment group was displayed using a Kaplan-Meier curve. The date of last dose of study medication was considered as the event date and also as the censoring date for those patients who did not discontinue treatment earl
Time Frame: 56 weeks
Population: The Safety set consisted of all patients that received at least one dose of study medication and had at least one post-baseline safety assessment. Patients were analyzed according to treatment received.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od
Number analyzed (Participants) | 204 | 204 | 206
Days | 384.0 (0.164) [384.0 to NA] — NA- Not estimable | NA (0.164) [NA to NA] — NA- Not estimable | NA (0.166) [NA to NA] — NA- Not estimable

3. Secondary Outcome: Change From Baseline in Pre-dose Trough FEV1
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FEV1 was defined as the average of the pre-dose FEV1 measured at -45 minutes (min) and -15 min at day 1. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline FEV1 measurements, smoking status at baseline, baseline inhaled corticosteroid (ICS) use, region, baseline FEV1 * visit interaction, and visit, treatment * visit interaction.
Time Frame: Day 29, 57,, 85, 141, 197, 253, 309 and 365
Population: The Full Analysis set (FAS) included all randomized patients who received at least one dose of study medication. Participants, who had both baseline and week 52 values, were included in the analysis. Patients were analyzed according to the treatment to which they were randomized.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od
Number analyzed (Participants) | 192 | 196 | 199
Liters
  Day 29 | 0.164 (0.0144) | 0.194 (0.0143) | 0.109 (0.0143)
  Day 57 | 0.178 (0.0151) | 0.199 (0.0149) | 0.107 (0.0149)
  Day 85 | 0.166 (0.0158) | 0.201 (0.0157) | 0.095 (0.0157)
  Day 141 | 0.174 (0.0173) | 0.198 (0.0170) | 0.087 (0.0171)
  Day 197 | 0.138 (0.0167) | 0.181 (0.0165) | 0.079 (0.0166)
  Day 253 | 0.142 (0.0168) | 0.153 (0.0165) | 0.074 (0.0167)
  Day 309 | 0.096 (0.0162) | 0.123 (0.0161) | 0.050 (0.0162)
  Day 365 | 0.116 (0.0169) | 0.116 (0.0167) | 0.037 (0.0169)

4. Secondary Outcome: Change From Baseline in 1 Hour Post-dose FEV1 Measurements
Description: as for outcome 3
Time Frame: Day 1, 29, 57, 85, 141, 197, 253, 309, and 365
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od
Number analyzed (Participants) | 200 | 202 | 202
Liters
  Day 1 | 0.166 (0.0088) | 0.178 (0.0088) | 0.122 (0.0089)
  Day 29 | 0.257 (0.0152) | 0.287 (0.0151) | 0.173 (0.0151)
  Day 57 | 0.267 (0.0157) | 0.302 (0.0155) | 0.173 (0.0154)
  Day 85 | 0.269 (0.0164) | 0.301 (0.0162) | 0.170 (0.0162)
  Day 141 | 0.268 (0.0182) | 0.288 (0.0179) | 0.170 (0.0181)
  Day 197 | 0.229 (0.0178) | 0.278 (0.0175) | 0.157 (0.0177)
  Day 253 | 0.231 (0.0178) | 0.240 (0.0175) | 0.140 (0.0176)
  Day 309 | 0.199 (0.0170) | 0.222 (0.0169) | 0.125 (0.0170)
  Day 365 | 0.212 (0.0175) | 0.221 (0.0173) | 0.104 (0.0174)

5. Secondary Outcome: Change From Baseline in FVC Measurement at All Post-baseline Time Points
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards.
Time Frame: Day1, 29, 57, 85, 141, 197, 253, 309, and 365
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od
Number analyzed (Participants) | 200 | 202 | 202
Liters
  Day 1 | 0.316 (0.0201) | 0.349 (0.0200) | 0.248 (0.0203)
  Day 29 | 0.375 (0.0274) | 0.440 (0.0271) | 0.280 (0.0272)
  Day 57 | 0.390 (0.0274) | 0.439 (0.0271) | 0.279 (0.0271)
  Day 85 | 0.388 (0.0287) | 0.432 (0.0283) | 0.268 (0.0284)
  Day 141 | 0.382 (0.0297) | 0.403 (0.0292) | 0.235 (0.0295)
  Day 197 | 0.313 (0.0288) | 0.400 (0.0284) | 0.220 (0.0288)
  Day 253 | 0.310 (0.0303) | 0.365 (0.0298) | 0.205 (0.0301)
  Day 309 | 0.272 (0.0284) | 0.334 (0.0281) | 0.185 (0.0285)
  Day 365 | 0.312 (0.0286) | 0.323 (0.0282) | 0.139 (0.0286)

6. Secondary Outcome: Percentage of Participants Experiencing Moderate or Severe COPD Exacerbation
Description: Percentage of participants experiencing moderate or severe Chronic Obstructive Pulmonary Disease (COPD)
Time Frame: 52 weeks
Population: The Full Analysis set (FAS) included all randomized patients who received at least one dose of study medication. Participants, who had both baseline and week 52 values, were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od
Number analyzed (Participants) | 204 | 204 | 206
Percentage of participants | 23.5 | 24.9 | 27.0

7. Secondary Outcome: Change From Baseline in Mean Total Daily Symptom Scores
Description: The participant recorded symptom scores twice daily in the eDiary. The daily clinical symptoms included: cough, wheezing, shortness of breath, sputum volume, sputum color, and night time awakening. The range of scores for each assessment is 0 to 3 where 0 indications No symptom and 3 indicates a Severe symptom. The maximum daytime total score is 27 and the maximum nighttime total score is 27. The total daily symptom score is obtained by adding the scores for the morning and evening symptoms for each day. The maximum possible total daily score is 54. A negative change from baseline indicated improvement.
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od
Number analyzed (Participants) | 198 | 199 | 198
Score on a scale | -1.57 (0.133) | -1.56 (0.133) | -1.31 (0.135)

8. Secondary Outcome: Change From Baseline in the Daily Number of Puffs of Rescue Medication Over the 52 Week Period
Description: Participants completed an electronic diary (eDiary) twice daily at the same time in the morning and evening to record the number of puffs of rescue medication taken in the previous 12 hours.
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB149 75 ug od
Number analyzed (Participants) | 198 | 199 | 198
Number of puffs | -1.89 (0.164) | -1.62 (0.164) | -1.73 (0.166)

ADVERSE EVENTS:
Groups:
- QAB75: QVA149 27.5/25 μg capsules
Arm/Group | QVA149 27.5/12.5 ug Bid | QVA149 27.5/25 ug Bid | QAB75
Serious Adverse Events (participants affected / at risk) | 26/204 | 25/204 | 24/206
Other Adverse Events (participants affected / at risk) | 118/204 | 117/204 | 112/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 27.5/12.5 ug Bid (N=204) | QVA149 27.5/25 ug Bid (N=204) | QAB75 (N=206)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 0 | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 | 1 | 0
BRADYCARDIA (Cardiac disorders) | 0 | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 0 | 1 | 0
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0
SILENT MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0
ASPLENIA (Congenital, familial and genetic disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 0 | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
FACIAL PAIN (General disorders) | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1 | 0
H1N1 INFLUENZA (Infections and infestations) | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 0 | 1
MENINGITIS (Infections and infestations) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 4 | 1 | 2
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 0 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 2 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
BRAIN HERNIATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 0 | 1 | 0
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
BONE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
NON-SMALL CELL LUNG CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
BRAIN OEDEMA (Nervous system disorders) | 0 | 2 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 1 | 0
PANIC ATTACK (Psychiatric disorders) | 0 | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 10
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
AORTIC DISSECTION (Vascular disorders) | 1 | 0 | 1
HAEMATOMA (Vascular disorders) | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 27.5/12.5 ug Bid (N=204) | QVA149 27.5/25 ug Bid (N=204) | QAB75 (N=206)
CONSTIPATION (Gastrointestinal disorders) | 1 | 3 | 1
DIARRHOEA (Gastrointestinal disorders) | 5 | 2 | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 4 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 5 | 4
VOMITING (Gastrointestinal disorders) | 3 | 2 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 4 | 4
OEDEMA PERIPHERAL (General disorders) | 1 | 6 | 5
PYREXIA (General disorders) | 3 | 4 | 0
BRONCHITIS (Infections and infestations) | 2 | 7 | 8
INFLUENZA (Infections and infestations) | 1 | 2 | 4
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 | 4 | 6
NASOPHARYNGITIS (Infections and infestations) | 19 | 18 | 22
PHARYNGITIS (Infections and infestations) | 3 | 0 | 3
PNEUMONIA (Infections and infestations) | 5 | 3 | 1
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 3 | 2 | 6
RHINITIS (Infections and infestations) | 4 | 3 | 2
SINUSITIS (Infections and infestations) | 5 | 7 | 6
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 10 | 9
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 10 | 14 | 13
URINARY TRACT INFECTION (Infections and infestations) | 0 | 4 | 3
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 6 | 7
CONTUSION (Injury, poisoning and procedural complications) | 3 | 2 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 | 7 | 5
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
HEADACHE (Nervous system disorders) | 5 | 7 | 4
INSOMNIA (Psychiatric disorders) | 3 | 2 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 70 | 64 | 71
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 13 | 7
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
HYPERTENSION (Vascular disorders) | 5 | 10 | 4
HYPOTENSION (Vascular disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.